CLINICAL TRIAL: NCT03299569
Title: Establishing the Incidence of Tako-tsubo Cardiomyopathy in Scotland - the STARR Study
Brief Title: Establishing the Incidence of Tako-tsubo Cardiomyopathy in Scotland
Acronym: STARR
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Tayside (Other Government); NHS Lothian (Other Government); NHS Highlands (Other); NHS Ayrshire and Arran (Other); Golden Jubilee National Hospital (Other Government); NHS Greater Glasgow and Clyde (Other); NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/LO/1059
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Takotsubo Cardiomyopathy; Myocardial Infarction
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Takotsubo cardiomyopathy: All patients diagnosed with Takotsubo cardiomyopathy in Scotland since 2010.
- Myocardial Infarction: An equal number of myocardial infarction patients in NHS Grampian since 2010.

SUMMARY:
Acute stress-induced (Takotsubo cardiomyopathy) presents like a heart attack and is triggered by intense emotional or physical stress. Although coronary arteries are unobstructed, it has been suggested that the risk of death is similar to a myocardial infarction. The purpose of the STARR study is to identify all cases of Takotsubo in Scotland since 2010 and assess its epidemiology and outcomes.

DETAILED DESCRIPTION:
Public Health Scotland will identify all patients centrally coded under codes I42.8 (Other cardiomyopathies), I42.9 (Cardiomyopathy, unspecified) and I51.8 (Other ill-defined heart diseases), using the Community Health Index (CHI) numbers from January 2010. All identified CHI numbers will be thereafter cross-checked with their clinical data at participating health boards to confirm a diagnosis of takotsubo cardiomyopathy and a registry of all confirmed Takotsubo cases will be established.

Clinical data will be collected for all Takotsubo patients retrospectively and prospectively. This will be compared to two contemporaneous gender and age matched control populations:

1. a cohort of randomly selected individuals from the Scottish general population supplied by Public Health Scotland
2. patients with myocardial infarction (extracted through collaboration with, the High-STEACS investigators, NCT01852123).

Electronic data linkage will be performed by Public Health Scotland to assess outcomes, prescribing and scores of prediction.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with Takotsubo cardiomyopathy

Exclusion Criteria:

* NA

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Takotsubo cardiomyopathy in Scotland since 2010
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-07-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality and morbidity of takotsubo syndrome | 13 years
  To use a nation-wide cohort (and matched national-wide control populations) to establish the all-cause mortality and consequent all cause hospitalisation rates

SECONDARY OUTCOMES:
Specific causes of mortality and morbidity of takotsubo syndrome | 13 years
  To use a nation-wide cohort (and matched national-wide control populations) to establish the specific causes of mortality and morbidities requiring subsequent hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, MD, MRCP, Principal Investigator — University of Aberdeen
Locations (1):
- Cardiac Research Office, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad A, Lerman A, Rihal CS. Apical ballooning syndrome (Tako-Tsubo or stress cardiomyopathy): a mimic of acute myocardial infarction. Am Heart J. 2008 Mar;155(3):408-17. doi: 10.1016/j.ahj.2007.11.008. Epub 2008 Jan 31. PMID 18294473
- [Background] Templin C, Ghadri JR, Diekmann J, Napp LC, Bataiosu DR, Jaguszewski M, Cammann VL, Sarcon A, Geyer V, Neumann CA, Seifert B, Hellermann J, Schwyzer M, Eisenhardt K, Jenewein J, Franke J, Katus HA, Burgdorf C, Schunkert H, Moeller C, Thiele H, Bauersachs J, Tschope C, Schultheiss HP, Laney CA, Rajan L, Michels G, Pfister R, Ukena C, Bohm M, Erbel R, Cuneo A, Kuck KH, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Cuculi F, Banning A, Fischer TA, Vasankari T, Airaksinen KE, Fijalkowski M, Rynkiewicz A, Pawlak M, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Franz WM, Empen K, Felix SB, Delmas C, Lairez O, Erne P, Bax JJ, Ford I, Ruschitzka F, Prasad A, Luscher TF. Clinical Features and Outcomes of Takotsubo (Stress) Cardiomyopathy. N Engl J Med. 2015 Sep 3;373(10):929-38. doi: 10.1056/NEJMoa1406761. PMID 26332547
- [Background] Elesber AA, Prasad A, Lennon RJ, Wright RS, Lerman A, Rihal CS. Four-year recurrence rate and prognosis of the apical ballooning syndrome. J Am Coll Cardiol. 2007 Jul 31;50(5):448-52. doi: 10.1016/j.jacc.2007.03.050. Epub 2007 Jul 16. PMID 17662398
- [Background] Sy F, Basraon J, Zheng H, Singh M, Richina J, Ambrose JA. Frequency of Takotsubo cardiomyopathy in postmenopausal women presenting with an acute coronary syndrome. Am J Cardiol. 2013 Aug 15;112(4):479-82. doi: 10.1016/j.amjcard.2013.04.010. Epub 2013 May 16. PMID 23683950
- [Background] Wittstein IS, Thiemann DR, Lima JA, Baughman KL, Schulman SP, Gerstenblith G, Wu KC, Rade JJ, Bivalacqua TJ, Champion HC. Neurohumoral features of myocardial stunning due to sudden emotional stress. N Engl J Med. 2005 Feb 10;352(6):539-48. doi: 10.1056/NEJMoa043046. PMID 15703419
- [Background] Dawson DK, Neil CJ, Henning A, Cameron D, Jagpal B, Bruce M, Horowitz J, Frenneaux MP. Tako-Tsubo Cardiomyopathy: A Heart Stressed Out of Energy? JACC Cardiovasc Imaging. 2015 Aug;8(8):985-7. doi: 10.1016/j.jcmg.2014.10.004. Epub 2014 Nov 1. No abstract available. PMID 25499134
- [Background] Neil C, Nguyen TH, Kucia A, Crouch B, Sverdlov A, Chirkov Y, Mahadavan G, Selvanayagam J, Dawson D, Beltrame J, Zeitz C, Unger S, Redpath T, Frenneaux M, Horowitz J. Slowly resolving global myocardial inflammation/oedema in Tako-Tsubo cardiomyopathy: evidence from T2-weighted cardiac MRI. Heart. 2012 Sep;98(17):1278-84. doi: 10.1136/heartjnl-2011-301481. Epub 2012 Jul 11. PMID 22791656
- [Background] Madhavan M, Borlaug BA, Lerman A, Rihal CS, Prasad A. Stress hormone and circulating biomarker profile of apical ballooning syndrome (Takotsubo cardiomyopathy): insights into the clinical significance of B-type natriuretic peptide and troponin levels. Heart. 2009 Sep;95(17):1436-41. doi: 10.1136/hrt.2009.170399. Epub 2009 May 24. PMID 19468013
- [Background] Summers MR, Lennon RJ, Prasad A. Pre-morbid psychiatric and cardiovascular diseases in apical ballooning syndrome (tako-tsubo/stress-induced cardiomyopathy): potential pre-disposing factors? J Am Coll Cardiol. 2010 Feb 16;55(7):700-1. doi: 10.1016/j.jacc.2009.10.031. No abstract available. PMID 20170799
- [Background] Cross-Disorder Group of the Psychiatric Genomics Consortium. Identification of risk loci with shared effects on five major psychiatric disorders: a genome-wide analysis. Lancet. 2013 Apr 20;381(9875):1371-1379. doi: 10.1016/S0140-6736(12)62129-1. Epub 2013 Feb 28. PMID 23453885
- [Background] Arbustini E, Narula N, Dec GW, Reddy KS, Greenberg B, Kushwaha S, Marwick T, Pinney S, Bellazzi R, Favalli V, Kramer C, Roberts R, Zoghbi WA, Bonow R, Tavazzi L, Fuster V, Narula J. Reply: The MOGE(S) classification for a phenotype-genotype nomenclature of cardiomyopathy: more questions than answers? J Am Coll Cardiol. 2014 Jun 17;63(23):2584-2586. doi: 10.1016/j.jacc.2014.03.028. Epub 2014 Apr 23. No abstract available. PMID 24768880
- [Background] Chen X, Lee G, Maher BS, Fanous AH, Chen J, Zhao Z, Guo A, van den Oord E, Sullivan PF, Shi J, Levinson DF, Gejman PV, Sanders A, Duan J, Owen MJ, Craddock NJ, O'Donovan MC, Blackman J, Lewis D, Kirov GK, Qin W, Schwab S, Wildenauer D, Chowdari K, Nimgaonkar V, Straub RE, Weinberger DR, O'Neill FA, Walsh D, Bronstein M, Darvasi A, Lencz T, Malhotra AK, Rujescu D, Giegling I, Werge T, Hansen T, Ingason A, Noethen MM, Rietschel M, Cichon S, Djurovic S, Andreassen OA, Cantor RM, Ophoff R, Corvin A, Morris DW, Gill M, Pato CN, Pato MT, Macedo A, Gurling HM, McQuillin A, Pimm J, Hultman C, Lichtenstein P, Sklar P, Purcell SM, Scolnick E, St Clair D, Blackwood DH, Kendler KS; GROUP investigators; International Schizophrenia Consortium. GWA study data mining and independent replication identify cardiomyopathy-associated 5 (CMYA5) as a risk gene for schizophrenia. Mol Psychiatry. 2011 Nov;16(11):1117-29. doi: 10.1038/mp.2010.96. Epub 2010 Sep 14. PMID 20838396
- [Background] Ashbrook DG, Williams RW, Lu L, Hager R. A cross-species genetic analysis identifies candidate genes for mouse anxiety and human bipolar disorder. Front Behav Neurosci. 2015 Jul 1;9:171. doi: 10.3389/fnbeh.2015.00171. eCollection 2015. PMID 26190982
- [Background] McCalmon SA, Desjardins DM, Ahmad S, Davidoff KS, Snyder CM, Sato K, Ohashi K, Kielbasa OM, Mathew M, Ewen EP, Walsh K, Gavras H, Naya FJ. Modulation of angiotensin II-mediated cardiac remodeling by the MEF2A target gene Xirp2. Circ Res. 2010 Mar 19;106(5):952-60. doi: 10.1161/CIRCRESAHA.109.209007. Epub 2010 Jan 21. PMID 20093629
- [Background] Pison L, De Vusser P, Mullens W. Apical ballooning in relatives. Heart. 2004 Dec;90(12):e67. doi: 10.1136/hrt.2004.046813. PMID 15547001
- [Background] Kumar G, Holmes DR Jr, Prasad A. "Familial" apical ballooning syndrome (Takotsubo cardiomyopathy). Int J Cardiol. 2010 Oct 29;144(3):444-5. doi: 10.1016/j.ijcard.2009.03.078. Epub 2009 Apr 17. PMID 19375184
- [Background] Sharkey SW, Lips DL, Pink VR, Maron BJ. Daughter-mother tako-tsubo cardiomyopathy. Am J Cardiol. 2013 Jul 1;112(1):137-8. doi: 10.1016/j.amjcard.2013.02.063. Epub 2013 Apr 2. PMID 23561588
- [Background] Caretta G, Robba D, Vizzardi E, Bonadei I, Raddino R, Metra M. Tako-tsubo cardiomyopathy in two sisters: a chance finding or familial predisposition? Clin Res Cardiol. 2015 Jul;104(7):614-6. doi: 10.1007/s00392-015-0837-0. Epub 2015 Mar 6. No abstract available. PMID 25743177